CLINICAL TRIAL: NCT02049801
Title: A Phase I Study of MEK Inhibitor MEK162 Combined With Idarubicin and Cytarabine Induction in Patients With Relapsed/Refractory RAS-Mutated Acute Myeloid Leukemia
Brief Title: MEK Inhibitor MEK162, Idarubicin, and Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: logistics
Sponsor: Bruno C. Medeiros (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Bruno C. Medeiros, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-29150; NCI-2014-00169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMAML0030 (Other: Stanford University Hospitals and Clinics)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (MEK inhibitor, MEK162, idarubicin, cytarabine) (Experimental): INDUCTION THERAPY: Patients receive MEK inhibitor MEK162 PO BID on days -4 to -1 and days 5-18, cytarabine IV continuously over 24 hours on days 1-4, and idarubicin IV over 1 hour on days 1-3. Patients may receive a second course of induction at the discretion of the principal investigator.
  POST-REMISSION THERAPY: Patients receive cytarabine IV continuously over 24 hours on days 1-3, idarubicin IV over 1 hour on days 1 and 2, and MEK inhibitor MEK 162 PO BID on days 4-17. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: MEK inhibitor MEK162; Drug: idarubicin; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: MEK inhibitor MEK162 — Given PO
  Other Names: ARRY-162; ARRY-438162
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the MEK inhibitor MEK162 to see if it is safe in patients when combined with idarubicin and cytarabine. MEK inhibitor MEK162 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving MEK inhibitor MEK162, cytarabine, and idarubicin may be an effective treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine maximum tolerated dose (MTD) of MEK162 (MEK inhibitor MEK162) in patients with RAS-mutated acute myeloid leukemia (AML) when combined with sequential induction chemotherapy (3+4) as measured by development of grade 3-4 dose-limiting toxicities (DLT).

SECONDARY OBJECTIVES:

I. Analyze downstream inhibition of RAS signaling following therapy with single-agent MEK162 with exploratory pharmacodynamics (PD) studies.

II. Perform preliminary efficacy analysis of combination of MEK162 and induction chemotherapy (3+4) in patients with RAS-mutated AML by measuring complete remission rate, 2-year overall survival, and duration of response.

OUTLINE:

INDUCTION THERAPY: Patients receive MEK inhibitor MEK162 orally (PO) twice daily (BID) on days -4 to -1 and days 5-18, cytarabine intravenously (IV) continuously over 24 hours on days 1-4, and idarubicin IV over 1 hour on days 1-3. Patients may receive a second course of induction at the discretion of the principal investigator.

POST-REMISSION THERAPY: Patients receive cytarabine IV continuously over 24 hours on days 1-3, idarubicin IV over 1 hour on days 1 and 2, and MEK inhibitor MEK 162 PO BID on days 4-17. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Prior morphological diagnosis of AML other than acute promyelocytic leukemia according to the 2001 World Health Organization (WHO) diagnostic criteria; patients with biphenotypic, RAS-mutated acute leukemia are also eligible
* Requiring salvage chemotherapy for persistent/refractory or relapsed disease after at least one course of conventional chemotherapy, e.g. with "7+3", as defined by persistence of >= 20% myeloid blasts on bone marrow aspirate or peripheral blood smear; a bone marrow biopsy is not routinely required, but should be obtained if the aspirate is dilute, hypocellular, or inaspirable; outside bone marrow examinations performed within the stipulated time period are acceptable for screening as long as the slides are reviewed at the study institution; flow cytometric analysis of the bone marrow aspirate should be performed according to institutional practice guidelines
* Confirmed RAS mutation (NRAS or KRAS) or confirmed PTPN11 mutation, measured on peripheral blood or bone marrow aspirate as part of screening prior to study enrollment; mutation status must be confirmed within 45 days of initiation of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (ULN)
* Serum bilirubin =< 2 times ULN
* Serum creatinine =< 1.5 mg/dl and/or creatinine clearance >= 50 mL/min
* Ejection fraction >= 50% by echocardiogram
* Corrected QT (QTc) interval =< 480 ms
* Ability to take oral medications
* Ability to understand and the willingness to sign a written informed consent document
* Ability to undergo standard induction chemotherapy
* Ability to adhere to the study visit schedule and other protocol requirements
* Life expectancy of greater than 2 months
* Negative serum beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) performed locally within 72 hrs prior to first dose

Exclusion Criteria:

* Concomitant treatment with other anti-neoplastic agents, with the exception of hydroxyurea
* Anti-neoplastic treatment less than 14 days prior to enrollment, with the exceptions of hydroxyurea or, in the case of a patient with primary refractory AML, prior induction chemotherapy
* Prior therapy with a MEK inhibitor
* Uncontrolled opportunistic infection or treatment for opportunistic infection within 4 weeks of first day of study drug dosing
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MEK162, anthracycline, or cytarabine
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of MEK162 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Previous or concurrent malignancy with the following exceptions:

  * Carcinoma in situ
  * Adequately treated skin basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
  * In situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to the study
  * A primary malignancy which has been completely resected and in complete remission for >= 5 years
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting [CABG], coronary angioplasty, or stenting) < 6 months prior to screening
  * Symptomatic chronic heart failure
  * Evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia
* Uncontrolled arterial hypertension despite appropriate medical therapy
* Patients who have neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Known confirmed diagnosis of human immunodeficiency virus (HIV) infection or active viral hepatitis (hepatitis B or hepatitis C)
* Any surgical procedure, excluding central venous catheter placement, bone marrow biopsy, lumbar puncture, or other minor procedures (e.g., skin biopsy) within 14 days of day 1; patients who have undergone major surgery =< 21 days prior to starting study drug or who have not recovered from side effects of such procedure are ineligible for the study
* Pregnant or nursing (lactating) women confirmed by a positive hCG laboratory test

  * Women of child-bearing potential unless they are using highly effective methods of contraception throughout the study and for 30 days after study drug discontinuation
* Sexually active males unless they use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Unwillingness or inability to comply with the protocol
* Known active leukemia of the central nervous system
* Known history of Gilbert's syndrome
* History or current evidence of retinal pigment epithelial detachment (RPED), retinal vein occlusion (RVO), or predisposing factors to RPED or RVO (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, hyperviscosity or hypercoagulability syndromes)
* History of retinal degenerative disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02-04 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
MTD of MEK inhibitor MEK162 in combination with chemotherapy, defined as the dose associated with a dose-limiting toxicity rate of 35% assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | 28 days
  Dose limiting toxicities will be tabulated by dose, severity and major organ system.

SECONDARY OUTCOMES:
Pharmacodynamic analysis of downstream inhibition of RAS signaling following therapy with single-agent MEK inhibitor MEK162 | Day -4, -1, and 18
  Pharmacodynamic correlative data will be summarized with medians and ranges for each dose group. If there are a sufficient number of patients assigned to both doses, the medians will be compared with a Wilcoxon Rank Sum test.
Complete remission rate, defined as bone marrow biopsy demonstrating < 5% blasts and recovery of peripheral blood counts after induction chemotherapy | Up to day 19
  The proportion of patients who achieve complete remission will be estimated overall with an exact 95% confidence interval; for descriptive purpose the same proportion at each dose will similarly described.
Overall survival | Time of study entry to the time of death from any cause, assessed at 2 years
  The proportion of patients who achieve 2-year overall survival will be estimated overall with an exact 95% confidence interval; for descriptive purpose the same proportion at each dose will similarly described.
Duration of response | Time of complete response to biopsy-documented recurrence of disease, assessed up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno de Medeiros, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No